CLINICAL TRIAL: NCT03312400
Title: Low Dose Danazol for the Treatment of Telomere Related Diseases
Brief Title: Low-Dose Danazol for the Treatment of Telomere Related Diseases
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 180004; 18-H-0004
Record Dates: First submitted 2017-10-14; First posted 2017-10-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12-09

CONDITIONS: Telomere Disease
Keywords: Telomeres; Aplastic Anemia; Pulmonary Fibrosis; Androgens; Hepatic Fibrosis
MeSH Terms: conditions — Anemia, Aplastic; Pulmonary Fibrosis; Liver Cirrhosis | interventions — Danazol

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 200 mg Arm (Active Comparator): 100 mg twice a day
  Interventions: Drug: Danazol
- 400 mg Arm (Active Comparator): 200 mg twice a day
  Interventions: Drug: Danazol

INTERVENTIONS:
Drug: Danazol — Adult: 200 mg daily versus 400 mg daily Pediatric: 4 mg/kg/day divided in twice daily dose (max 400 mg daily) for 6 months or 2 mg/kg/day divided in twice daily dose (max 200 mg daily) for 6 months.

SUMMARY:
Background:

DNA is a structure in the body. It contains data about how the body develops and works. Telomeres are found on the end of chromosomes in DNA. Some people with short telomeres or other gene changes can develop diseases of the bone marrow, lung, and liver. Researchers want to see if low doses of the hormone drug danazol can help.

Objective:

To study the safety and effect of low dose danazol.

Eligibility:

People ages 3 and older with a telomere disease who have either very short telomeres and a specific gene change. They must also show signs of aplastic anemia, lung, or liver disease.

Design:

Participants will be screened in another protocol.

Participants will have:

* Medical history
* Physical exam
* Blood tests
* Lung exam. They will breathe into an instrument that records the amount and rate of air breathed in and out over a period of time.

  6-minute walking test.
* Abdominal ultrasound and liver scan. These tests use sound waves to measure the fibrosis in the liver.

Some participants will have:

* Pregnancy test
* Small sample of the liver removed
* Bone marrow biopsy. The bone will be numbed and a small needle will take a sample of the marrow.

All participants will have hormone levels checked.

All child participants will see a pediatric endocrinologist. Children may need to have a hand x-ray.

We will monitor patients for 6 months before starting danazol.

Participants will take danazol by mouth twice a day for 1 year.

Participants must return to the clinic at 6 months and 12 months while on danazol and 6 months after stopping it. They will have blood and urine tests, a lung exam, abdominal ultrasound, and liver scan.

DETAILED DESCRIPTION:
Telomere disease is caused by accelerated telomere attrition and results in multi-organ dysfunction. Telomeres are nucleotide repeats of non-coding DNA at the end of the chromosomes which function as protective caps to prevent erosion of genomic DNA during cell division and to protect chromosomes from recognition as single stranded DNA. Telomeric DNA is elongated by the telomerase complex, which is comprised of a reverse transcriptase catalytic subunit (encoded by TERT), an RNA template (encoded by TERC) and associated proteins.

Telomerase activity is crucial in maintaining telomere length in cells with a high proliferative capacity, such as hematopoietic stem cells (HSCs) and lymphocytes. Presentation of telomeropathies can vary from severe aplastic anemia (SAA) and dyskeratosis congenital (DKC) early in childhood, to pulmonary or hepatic fibrosis later in life. There is no standard of care for the treatment of telomere disease.

Considerable evidence suggests that sex hormones regulate telomerase. Calado et al. demonstrated that human lymphocytes and CD34+ hematopoietic cells up regulate both TERT gene expression and telomerase enzymatic activity in response to androgens in vitro. A recent observational cohort study demonstrated hematologic response in 14 of 16 pediatric patients with DKC treated with androgens. In a prospective trial from our Branch, Townsley et al demonstrated that patients with telomere diseases who were treated with the synthetic sex hormone danazol showed telomere elongation, and hematologic response were seen in 79% of patients after only three months of treatment. This study used the highest dose of danazol, 800 mg daily, and known adverse effects, such as elevated liver enzyme levels and muscle cramps, occurred in 41% and 33% of patients, respectively. Overall the treatment was well tolerated, but some patients did require dose reduction. After 27 patients were enrolled, the study was halted early, because telomere attrition was reduced in all 12 patients who could be evaluated for the primary endpoint. Because of the limited power, we were unable to draw definitive conclusions regarding further clinical effect of danazol but stabilization or improvement was observed in a few cases in other organ function, measured by DLCO for pulmonary fibrosis and Fibroscan for cirrhosis.

We now propose a phase II study designed to determine the efficacy of low dose danazol in decreasing the rate of telomere attrition in subjects with a short age-adjusted telomere length. The secondary aim is to determine the clinical effect of this therapy in conditions that are related to short telomeres, to include cytopenia(s), pulmonary fibrosis, and/or hepatic fibrosis.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Age-adjusted telomere length less than or equal to the first percentile by flow-FISH method. In patients with a known pathogenic or likely pathogenic mutation in a telomere maintenance gene, age adjusted telomere length less than or equal to the 10th percentile is sufficient.
  2. A mutation in telomere maintenance genes (TERT, TERC, DKC1, TINF2, NHP2, NOP10, WRAP53, TERF2, PARN, RTEL1, ACD, CTC1, USB1) as tested in a CLIA (or international equivalent) certified laboratory
  3. Age greater than or equal to 3 years
  4. Weight greater than or equal to 12 Kg

     AND
  5. At least one of the following criteria:

     1. Anemia with a hemoglobin less than or equal to 10 g/dL without red blood cell transfusion
     2. Thrombocytopenia with a platelet count less than or equal to 50,000/microliter without transfusion
     3. Neutropenia with an absolute neutrophil count less than or equal to 1,000/ microliter

     OR

     Pulmonary fibrosis diagnosed by either a lung biopsy or computed tomography scan of the chest according to guidelines from the American Thoracic Society and European Respiratory Society.

     OR
  6. Hepatic fibrosis diagnosed by Transient Elastography by Fibroscan value greater than 10 kpa or US evidence of cirrhotic liver or splenomegaly, or transjugular liver biopsy demonstrating fibrosis.

EXCLUSION CRITERIA:

1. Patients on androgen hormones to include testosterone or high dose estrogen (estradiol 0.5 mg/day or greater) for the12 months prior to enrollment
2. Patients with active thrombosis or thromboembolic disease and history of such events, undiagnosed abnormal genital bleeding, porphyria, androgendependent tumor, or prostatic hypertrophy
3. Patients with pulmonary fibrosis who are receiving anti-fibrotic drug treatment, such as pirfenidone or nintedanib unless stable on anti-fibrotic drug for at least 6 months prior to starting on danazol as demonstrated by PFTs.
4. Patients with active hepatitis B or C
5. Patients who have received a bone marrow transplant
6. Patient with other hereditary bone marrow failure syndromes such as Fanconi anemia or Diamond Blackfan anemia
7. Patients with infections not adequately responding to appropriate therapy
8. Current pregnancy, or unwillingness to take oral contraceptives or use the barrier methods of birth control or practice abstinence to refrain from pregnancy if of childbearing potential during the course of the study
9. Lactating women, due to the potentially harmful effects on the nursing child
10. Patients with cancer who are actively receiving systemic chemotherapeutic treatment or who take drugs with hematological effects
11. Patients with decompensated liver disease to include persistent ascites, encephalopathy, variceal hemorrhage, or MELD score of 10 or greater
12. Inability to understand the investigational nature of the study or to give informed consent or without a legally authorized representative or surrogate that can provide informed consent
13. Inability to swallow a capsule

Ages: 3 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-02-08 (Actual); Primary Completion 2026-04-29 (Estimated); Study Completion 2027-10-29 (Estimated)

PRIMARY OUTCOMES:
Reduction of telomere attrition rate | Over 6 months
  Reduction of telomere attrition rate (decreased rate of telomere attrition by 50%, as compared to the baseline rate)

SECONDARY OUTCOMES:
Toxicities associated with low dose danazol use | During 12 months of treatment
Progression of pulmonary function testing | After 6 and 12 months of treatment
Progression of fibroscan and transient elastography by ARFI | After 6 and 12 months of treatment
Hematologic response | After 6 and 12 months of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Emma M Groarke, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known

REFERENCES:
- [Background] Calado RT, Yewdell WT, Wilkerson KL, Regal JA, Kajigaya S, Stratakis CA, Young NS. Sex hormones, acting on the TERT gene, increase telomerase activity in human primary hematopoietic cells. Blood. 2009 Sep 10;114(11):2236-43. doi: 10.1182/blood-2008-09-178871. Epub 2009 Jun 26. PMID 19561322
- [Background] Townsley DM, Dumitriu B, Liu D, Biancotto A, Weinstein B, Chen C, Hardy N, Mihalek AD, Lingala S, Kim YJ, Yao J, Jones E, Gochuico BR, Heller T, Wu CO, Calado RT, Scheinberg P, Young NS. Danazol Treatment for Telomere Diseases. N Engl J Med. 2016 May 19;374(20):1922-31. doi: 10.1056/NEJMoa1515319. PMID 27192671
- [Background] Khincha PP, Wentzensen IM, Giri N, Alter BP, Savage SA. Response to androgen therapy in patients with dyskeratosis congenita. Br J Haematol. 2014 May;165(3):349-57. doi: 10.1111/bjh.12748. Epub 2014 Feb 12. PMID 24666134
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2018-H-0004.html